CLINICAL TRIAL: NCT03976154
Title: The Effects of Fixation Technique On Thoracic Epidural Catheter Displacement: A Single-Center Randomized Controlled Trial
Brief Title: Effects of Fixation Technique On Thoracic Epidural Catheter Displacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Meier, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122914
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Thoracic Epidural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dermabond (Experimental): Catheter fixation will be performed after appropriate placement of a thoracic epidural with Dermabond. The investigator performing the thoracic epidural will distribute the Dermabond at the catheter insertion site in a space no greater than a 2 cm circle around the site. Once the Dermabond is allowed to dry, mastisol will be applied to the surrounding skin and a clear Tegaderm dressing will be used to cover the catheter. Catheter depth at the skin will be recorded at that time. An Epidural catheter infusion pump with 1/8thpercent Bupivacaine and 2mcg/ml Fentanyl will be attached to the catheter and started by the primary anesthesia with a goal rate of 6ml/hr.
  Interventions: Other: Thoracic Epidural Catheter Fixation Techniques
- Mastisol (Active Comparator): Catheter fixation will be performed after appropriate placement of a thoracic epidural with Mastisol spray. The investigator performing the epidural placement will distribute Mastisol spray both in close proximity to the catheter insertion site as well as around the insertion site. Once the Mastisol is allowed to dry, a clear Tegaderm dressing will be used to cover the catheter. Catheter depth at the skin will be recorded at that time. An Epidural catheter infusion pump with 1/8thpercent Bupivacaine and 2mcg/ml Fentanyl will be attached to the catheter and started by the primary anesthesia team with a goal rate of 6ml/hr.
  Interventions: Other: Thoracic Epidural Catheter Fixation Techniques
- Grip-lock (Active Comparator): Catheter fixation will be performed after appropriate placement of a thoracic epidural with a Grip-Lok fixation bandage. The investigator performing the epidural placement will place the fixation bandage one centimeter caudal from the insertion site. Mastisol will be applied to the surrounding skin and a clear Tegaderm will then be used to cover the catheter. Catheter depth at the skin will be recorded at that time. An Epidural catheter infusion pump with 1/8thpercent Bupivacaine and 2mcg/ml Fentanyl will be attached to the catheter and started by the primary anesthesia team in the operating room with a goal rate of 6ml/hr.
  Interventions: Other: Thoracic Epidural Catheter Fixation Techniques

INTERVENTIONS:
Other: Thoracic Epidural Catheter Fixation Techniques — All thoracic epidurals will be placed by a regional anesthesia resident or fellow under the direct supervision of an attending anesthesiologist using a standard epidural kit and in the paramedian approach.
  Epidural placement will occur preoperatively in the same manner as our current practice criterion. There will be no difference in placement of the epidural catheter between the control groups and the treatment group. After placement, catheters will be secured with either Dermabond, Mastisol, or a Grip-Lok fixation bandage, all with overlying Tegaderms.

SUMMARY:
The purpose of our study is to assess the effectiveness of Dermabond as a thoracic epidural fixation technique compared to both Mastisol and the Grip-Lok fixation bandage, two common, widely used techniques for epidural fixation.

ELIGIBILITY:
Inclusion Criteria:

* surgical patient
* receiving a thoracic epidural
* 18 years of age or older

Exclusion Criteria:

* Patient refusal
* allergy to adhesives or local anesthesia
* pregnancy
* contraindication to receiving an epidural including coagulopathy, infection, elevated ICP, or severe pre-existing neurologic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidural catheter displacement immediately after surgery | immediately after surgery in PACU
  Failure of epidural fixation as measured by catheter depth at the skin (to the nearest 0.5 cm
Epidural catheter displacement day 1 | 24 hours post-operative
  Failure of epidural fixation as measured by catheter depth at the skin (to the nearest 0.5 cm
Epidural catheter displacement day 2 | 48 hours post-operative
  Failure of epidural fixation as measured by catheter depth at the skin (to the nearest 0.5 cm
Epidural catheter displacement day 3 | 72 hours post-operative
  Failure of epidural fixation as measured by catheter depth at the skin (to the nearest 0.5 cm
Epidural catheter displacement day 4 | 96 hours post-operative
  Failure of epidural fixation as measured by catheter depth at the skin (to the nearest 0.5 cm
Epidural catheter displacement day 5 | 120 hours post-operative
  Failure of epidural fixation as measured by catheter depth at the skin (to the nearest 0.5 cm
Epidural catheter displacement day 6 | 144 hours post-operative
  Failure of epidural fixation as measured by catheter depth at the skin (to the nearest 0.5 cm
Epidural catheter displacement day 7 | 168 hours post-operative
  Failure of epidural fixation as measured by catheter depth at the skin (to the nearest 0.5 cm

SECONDARY OUTCOMES:
Leakage | immediately after surgery in PACU and daily until the patient is discharged up to post-operative day 7
  presence of any leakage from catheter fixation
Percent of patients with skin changes as measured by clinician subjective assessment | immediately after surgery in PACU and daily until the patient is discharged up to post-operative day 7
  The clinician will subjectively assess any skin changes including induration or erythema
Opioid consumption | daily up to 7 days post-operative
  Daily oral morphine equivalent totals

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No